CLINICAL TRIAL: NCT00105170
Title: A Phase I, Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Safety and Tolerability of hCBE-11, a Humanized Monoclonal Antibody, in Subjects With Advanced Solid Tumors
Brief Title: Safety and Tolerability of hCBE-11 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202-01
Record Dates: First submitted 2005-03-08; First posted 2005-03-09 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Tumors
Keywords: Monoclonal antibody; Advanced solid tumors; Tumors; hCBE-11
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: hCBE-11

SUMMARY:
This is a Phase I, open-label, dose-escalation study on subjects with advanced solid tumors. This is the first study of hCBE-11 in humans and is designed to determine the safety and how well patients tolerate this investigational drug. The study duration is two years with treatment visits occurring weekly for either 4 or 8 weeks, follow-up for 8 weeks and long-term follow-up contact every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory solid tumors not curable with standard therapy.
* At least one measurable lesion
* ECOG Performance Status less than or equal to 2
* Acceptable hematologic status
* Albumin greater than or equal to 2.5 g/dL
* Normal calculated glomerular filtration rate (GFR)
* Acceptable liver function

Exclusion Criteria:

* Uncontrolled cardiac disease, angina, congestive heart failure, or myocardial infarction within 6 months prior to Study Day
* Known history of hepatitis B or C, or HIV infection
* Clinically significant effusions, including pericardial, pleural, and ascites
* Serious non-malignant disease
* Central nervous system (CNS) metastatic involvement except where the disease has been successfully treated
* Investigational therapies within 4 weeks of Study Day 1
* Radiation therapy of tumors to be followed for this study
* Chemotherapy, biologic therapy, or major surgery other than diagnostic within 4 weeks prior to Study Day 1
* Current Grade 3 or 4 neurological toxicity
* Concurrent anti-neoplastic therapy and/or steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of hCBE-11 in advanced solid tumors | up to 2 years

SECONDARY OUTCOMES:
To define the recommended Phase II dose of hCBE-11 | up to 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Tucson, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Philadelphia, Pennsylvania